CLINICAL TRIAL: NCT01682473
Title: A Phase 1, Multi-Center, Open Label, Uncontrolled, Serial Cohort, Dose Escalation Study of the Safety, Tolerability, Pharmacokinetics and Efficacy of ZSTK474 in Japanese Patients With Advanced Solid Malignancies
Brief Title: A Study of ZSTK474 in Japanese Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zenyaku Kogyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZSTK474-201
Record Dates: First submitted 2012-09-04; First posted 2012-09-11 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Neoplasms
Keywords: PI3K inhibitor; clinical trial
MeSH Terms: conditions — Neoplasms | interventions — ZSTK474

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: 5/2 Dosing (Experimental): Subjects will receive oral ZSTK474 at a fixed once daily dose administered in 4-week (28-day) cycles of 5 days on drug and 2 days off drug.
  Interventions: Drug: ZSTK474
- Arm 2: 21/7 Dosing (Experimental): Subjects will receive oral ZSTK474 at a fixed once daily dose administered in 4-week (28-day) cycles of 21 days on drug and 7 days off drug.
  Interventions: Drug: ZSTK474

INTERVENTIONS:
Drug: ZSTK474 — Two arms, each with serial cohorts receiving escalating doses.

SUMMARY:
To evaluate the safety (adverse events and dose-limiting toxicity) of daily oral doses of ZSTK474 in patients with advanced solid malignancies.

DETAILED DESCRIPTION:
Open-label, uncontrolled, serial cohort, dose-escalation study evaluating two different dosing regimens (Arm 1: cycles of 5 days on drug and 2 days off drug), Arm 2: cycles of 21 days on drug and 7 days off drug).

ELIGIBILITY:
Inclusion Criteria:

* Japanese males or females >= 20 years old
* Advanced (metastatic or unresectable) solid tumor
* ECOG performance status score of 0 or 1 and expected survival >12 weeks
* Recovered from hematological toxicities of prior cancer therapies

Exclusion Criteria:

* Previous treatment with PI3K inhibitor
* Serious/significant illnesses or underlying conditions, including diabetes or hepatic renal or CV disease.
* Other investigational agent within previous 4 weeks
* Participating in another clinical study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09-20 (Actual); Primary Completion 2015-04-02 (Actual); Study Completion 2015-04-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities | 28 days

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax, tmax, t½, AUC) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Toshihiko Doi, MD, PhD, Principal Investigator — National Cancer Center Hospital East; Shunji Takahashi, MD, Principal Investigator — The Cancer Institute Hospital of JFCR
Locations (2):
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo